CLINICAL TRIAL: NCT03272386
Title: Verbal Instruction to Obtain Voluntary Pelvic Floor Muscle Contraction: Acceptability, Understanding and Best Instruction
Brief Title: Best Verbal Instruction to Obtain Voluntary Pelvic Floor Muscle Contraction
Status: Completed | Type: Observational
Sponsor: Pierre and Marie Curie University (Other)
Responsible Party: Principal Investigator, Gérard Amarenco, Head of Neuro-Urology department, Tenon hospital, Pierre and Marie Curie University
Other Study IDs: P. GREEN 01
Record Dates: First submitted 2017-08-16; First posted 2017-09-05 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: pelvic floor muscles; instruction; assessment; acceptability; understanding
MeSH Terms: conditions — Lower Urinary Tract Symptoms | interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational study: Observational study with patients over 18 years old, consulting for lower urinary tract symptoms in a tertiary center are included.
  Interventions: Other: Observational study

INTERVENTIONS:
Other: Observational study — Completing a questionnaire

SUMMARY:
The purpose of this study is to determine the best verbal instruction to obtain a PFMC and to evaluate the understanding and acceptability of the proposed instructions.

DETAILED DESCRIPTION:
Pelvic floor muscles contraction (PFMC) is usually recommended for evaluation and treatment of pelvic floor disorders.

In clinical practice, many patients fail to achieve a voluntary PFMC and only about one-third of women perform an ideal PFMC after brief written or verbal instruction. When no PFMC is elicited, it might be explained by an anatomical or neurological issue but also by a lack of understanding of the instructions and / or poor knowledge of the anatomy. Pelvic floor muscles (PFM) evaluation may depends on the method used to elicit and assess the contraction including verbal instructions. There is no current gold standard methodology for quantifying PFM strength and the verbal instructions used to elicit the PFMC are rarely reported in the studies. There is few specific works about the instructions. One recent study report that the pattern of urethral movement is influenced by the instructions used to teach activation of the PFM in men. Another study showed that some specific instructions are most effective in eliciting a correct PFMC in women.

Thus, an appropriate verbal instruction in terms of understanding, social and cultural acceptability, taking into account the anatomical knowledge of the patients, would probably allow a better evaluation of the PFM and even a better efficacy of pelvic floor training.

The purpose of this study is to determine the best verbal instruction to obtain a PFMC and to evaluate the understanding and acceptability of the proposed instructions.

This is a prospective observational study lead in two phases in the Neurourology Department of a University Hospital.

Phase 1: survey carry out the health professionals. Members of the scientific committees of national academic societies in neuro-urology, pelvi-perineology and pelvic-floor neurophysiology would be invited to answer a questionnaire by mail. It will include open questions about the most frequently verbal instructions used to elicit a PFMC. These instructions will be collected, analysed and selected for the second phase.

Phase 2: structured interviews with patients and with non-health professional subjects.

Patients and non-health professionals subjects will be invited to answer a 3-parts questionnaire based on the gender: (i) demographic, social and medical data; (ii) evaluation of the anatomical knowledge of the perineum with a picture of the perineum and a sagittal section of the pelvic area of the corresponding sex. In the third part (iii), the participants will assess the instructions selected in the first phase according to their understanding and their acceptability (good, intermediate, poor). They finally will have to choose the best instruction i.e. which seems to be the more suitable to obtain a PFMC.

Ethics: a local ethics committee approved this study. Since it is an observational study, the participant will have a newsletter.

ELIGIBILITY:
Inclusion Criteria:

* Follow in neuro-urology
* Lower urinary tract symptoms

Exclusion Criteria:

* Can't speak French

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients consulting in a tertiary center in neuro-urology.
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Description of the instructions used by the professionals | 1 day during the consultation
  Qualitative description of the instructions and selection of the most frequent instructions.

SECONDARY OUTCOMES:
Acceptability, understanding and selection of the best instruction by the subjects | 1 day during the consultation
  Description of the selected instructions by the subjects : their acceptability (poor / moderate / good), and understanding (poor / moderate / good) and the best instruction to obtain PFMC (among the selected instructions).

CONTACTS AND LOCATIONS:
Overall Officials: Gérard Amarenco, PhD, Principal Investigator — UPMC, Sorbonne Université, Univ Paris 6, service neuro-urologie, hôpital TENON, Paris
Locations (1):
- Department of neuro-urology, hôpital Tenon, Paris, France